CLINICAL TRIAL: NCT00791050
Title: To Examine the Effects on Patients Outcomes of Maintaining Body Core Temperature During CABGs With Thermowrap
Brief Title: Examine the Effects of Maintaining Body Core Temperature During CABGs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Luca Salvi, MD, IRCCS Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCMAneste002
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-10

CONDITIONS: Anesthesia; Hypothermia; Coronary Artery Bypass Grafting
Keywords: Hypothermia/complications/etiology; coronary artery bypass/adverse effects
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Thermo (Experimental)
  Interventions: Device: Allon Thermowrap. MTRE Advanced Technologies Ltd.
- 2 Control (No Intervention)

INTERVENTIONS:
Device: Allon Thermowrap. MTRE Advanced Technologies Ltd. — Thermowrap set at 37 °C before induction of anesthesia and maintained until initiation of CPB; during CPB set to "monitoring" and set again to 37 °C from rewarming during CPB to end of surgery.
  Arms: 1 Thermo

SUMMARY:
Although data on cardioprotective effects (as profile of troponin I)of perioperative maintenance of normothermia during CABGs are already known, little is known about the effects of maintaining normothermia on clinical outcomes of patients submitted to coronary surgery. Being acute renal failure (ARF) and atrial fibrillation (AF) the two most frequent complications of this surgery, this study compare as primary end point the rate of postoperative ARF and AF in two group of patients, one actively warmed with Thermowrap and the control group receiving standard institutional care.

ELIGIBILITY:
Inclusion Criteria:

* Isolated on pump CABGs
* Age 18 - 85
* Preoperative core temperature 36- 37.5 °C

Exclusion Criteria:

* History of fever in the last week
* Severe renal, hepatic,hematologic or pulmonary disease
* Chronic Atrial fibrillation
* History of acute MI in the last week
* Previous neurologic abnormalities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Rate of atrial fibrillation | First 48 postoperative hours
Rate of acute renal failure | First 48 postoperative hours

SECONDARY OUTCOMES:
Rate of Myocardial infarction and low output syndrome | First postoperative 48 hours
Rate of Type I neurological injury | First 48 postoperative hours
Total units of RBCs transfused | First 48 postoperative hours
Length of mechanical ventilation | First 48 postoperative hours
Rate of in-hospital mortality | 30 postoperative days
Intensive Care Unit length of stay | 30 postoperative days
Hospital length of stay | 30 postoperative days
Cardiac Troponin I (cTnI) curve | First postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luca Salvi, MD, Principal Investigator — Dept. of Anesthesia & ICU, IRCCS Centro Cardiologico Monzino. Milano, Italy
Locations (1):
- Dept. of Anesthesia & ICU, IRCCS Centro Cardiologico Monzino, Milan, Italy

REFERENCES:
- [Background] Nesher N, Zisman E, Wolf T, Sharony R, Bolotin G, David M, Uretzky G, Pizov R. Strict thermoregulation attenuates myocardial injury during coronary artery bypass graft surgery as reflected by reduced levels of cardiac-specific troponin I. Anesth Analg. 2003 Feb;96(2):328-35, table of contents. doi: 10.1097/00000539-200302000-00007. PMID 12538173